CLINICAL TRIAL: NCT05523973
Title: Effects of Lingual Endurance Exercise on Rehabilitation of Swallowing Impairment After Ischemic Stroke
Brief Title: Lingual Endurance Exercise in Treating Post-Stroke Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Brittany Krekeler, Assistant Professor, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0218; P2CHD101899 (NIH)
Record Dates: First submitted 2022-08-25; First posted 2022-09-01 (Actual); Results first posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Dysphagia, Oral Phase; Stroke, Ischemic
Keywords: swallowing; dysphagia; sub-acute stroke; tongue; exercise
MeSH Terms: conditions — Deglutition Disorders; Ischemic Stroke; Motor Activity

STUDY DESIGN:
Intervention Model Description: Some participants will practice only lingual endurance exercise 3 times a day, others will have a effortful swallow exercise to practice in place of their third session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lingual Endurance Training (Experimental): Participants will complete lingual endurance training 2-3 times a day. Half of the participants will also complete a session of effortful swallows with the device.
  Interventions: Other: Lingual Endurance Training

INTERVENTIONS:
Other: Lingual Endurance Training — Participants will participate in 3 training sessions per day for 8 weeks. Some participants will complete 3 sessions of lingual endurance exercise. For example, if the participant completed 100 repetitions during the baseline measurement, they would complete 75 repetitions during their exercise session. Other participants will complete effortful swallows during their 3rd training session. These participants will complete 30 swallows where they are instructed to press their tongue hard on the bulb and swallow their saliva.

SUMMARY:
Aim 1: Determine feasibility of lingual endurance training for individuals with persistent dysphagia after ischemic stroke. Primary outcome measures: % patient adherence (# of attempted repetitions/# prescribed repetitions) and % dose delivery (# of repetitions meeting goal/# prescribed repetitions). Aim 2: Determine preliminary efficacy of lingual endurance training on improving critical aspects of oropharyngeal swallowing (physiologic impairments, clearance of oropharyngeal residue, airway protection), functional oral intake, and patient reported swallowing quality of life in individuals with persistent dysphagia after ischemic stroke. Primary outcome measures: improvement on videofluoroscopic assessment of swallowing function using the gold standard Modified Barium Swallowing Impairment Profile (MBSImP) Overall Impression (OI) score and Functional Oral Intake Scale (FOIS) score. Secondary outcome measures: Analysis of Swallow Physiology, Events, Timing and Kinematics (ASPEKT); airway invasion - Penetration Aspiration Scale (PAS). Patient reported outcome measures: EAT-10 (Eating Assessment Tool) and the Swallowing Quality of Life Questionnaire (SWAL-QoL).

DETAILED DESCRIPTION:
Implications of Post-Stroke Dysphagia Dysphagia (swallowing impairment) after stroke is common, estimated to affect 78% of patients.1 Dysphagia results in additional negative consequences that complicate patient recovery and increase the risk of developing pulmonary complications (aspiration pneumonia) and may result in suboptimal nutrition. These comorbidities increase cost of care, up to $6,243 on average per patient, placing a burden not only on the individual, but also the healthcare system at large. The effects of dysphagia post-stroke extend beyond physical health concerns and increase the risk of depression, with devastating impacts on quality of life. Given these undesirable and dangerous health consequences, adequate assessment and treatment of swallowing impairments after stroke is a critical component of rehabilitation for this patient population.

Limitations to Current Treatment Approaches Current treatment approaches to alleviate dysphagia after stroke, especially in acute and sub-acute phases, have primarily focused on diet modification, compensatory posturing, and providing alternate access to hydration and nutrition. While the goal of these strategies is to improve swallow safety and avoid negative consequences of airway invasion, these techniques can be burdensome to the patient if implemented long-term. Additionally, these approaches do not target rehabilitation of swallowing function, but rather provide a somewhat temporary solution to what is, for many patients, a life-long issue. Available rehabilitative approaches to target improvements in function of oropharyngeal musculature during swallowing include both swallowing exercises (task-specific) and non-swallowing exercises (e.g. tongue exercise), which rely on the principles of transference to improve swallowing function. However, evidence is inconsistent regarding efficacy of these "exercise-based" interventions that target the oropharyngeal musculature, and the scientific validity of these trials varies greatly. Of these non-swallowing exercise approaches, lingual (tongue) exercise has been frequently studied and can be facilitated by medical devices which provide bio-feedback of lingual pressure generative capabilities to the patient and clinician. However, there is little to no evidence that lingual strengthening improves swallow physiology or functional outcomes in post-stroke dysphagia, and a majority of these previous studies lack use of standardized outcomes or randomized controlled trial procedures. Also, lingual strengthening may not induce biological changes to tongue muscle fiber size, as would be expected with a resistance-based exercise program. Despite these mixed findings, lingual strengthening is still routinely to treat post-stroke dysphagia. A major limitation of these current approaches is a sole focus on increasing muscular strength alone without consideration for other aspects of muscle physiology necessary for swallowing, such as endurance.

Lingual Endurance Training as an Alternative Approach In this preliminary study, we have proposed to examine the effects of lingual endurance training in individuals with dysphagia after stroke, as an alternative approach to traditional progressive lingual strength training, because this patient group is known to have specific deficits in lingual function after stroke. Both oral and pharyngeal tongue movements are essential for safe and efficient swallowing. Thus, exercise of the lingual musculature is a reasonable goal. However, swallowing is an endurance task; lingual pressures required for swallowing are submaximal, requiring repeated and sustained contraction over the course of a meal. Thus, targeting improvement in lingual endurance over strength alone may provide greater transferrable benefit to daily swallowing tasks. However, there are currently no randomized controlled trials investigating efficacy of lingual endurance training as a treatment for dysphagia in any patient population. As such, this proposed preliminary trial is essential to gathering the necessary pilot evidence regarding whether lingual endurance training is feasible and effective as an alternative approach to dysphagia rehabilitation for individuals with swallowing impairments after stroke. The long-term goal of this proposed work is to develop improved, evidence-based protocols for lingual exercise training for individuals with dysphagia after stroke. Ultimately, the results of this proposed pilot will be highly significant in creating movement towards more specific and evidence-based approaches for this unique patient group, who currently have very few rehabilitative options available. In this initial trial, we will assess if lingual endurance training will be feasible (Aim 1) and effective (Aim 2) for improving swallowing function in post-stroke dysphagia.

ELIGIBILITY:
Inclusion Criteria:

* ≥3 months since initial diagnosis ischemic, non-hemorrhagic stroke occurring in areas involving anterior or posterior circulation and affecting underlying cortical or subcortical structures (including brainstem)
* are safe to tolerate some oral intake required for assessment of swallowing function via Modified Barium Swallow Study
* able to follow 2-step commands
* English speaking. Participants will not be considered for inclusion if they meet any of the following screening exclusion criteria

Exclusion Criteria:

* a history of dysphagia prior to or after the stroke caused by any of the following conditions: gastrointestinal disease, traumatic brain injury, head and neck cancer, or a surgical procedure involving the pharynx or larynx
* a history of other neurological disease including traumatic brain injury, multiple sclerosis, Amyotrophic lateral sclerosis (ALS), Parkinson, or dementia
* Pregnant women
* Patients with a history of Temporomandibular joint dysfunction (TMJ) or Epilepsy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brittany Krekeler, PhD, Principal Investigator — University of Cincinnati, Department of Otolaryngology-Head and Neck Surgery
Locations (1):
- Medical Sciences Building, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martino R, Foley N, Bhogal S, Diamant N, Speechley M, Teasell R. Dysphagia after stroke: incidence, diagnosis, and pulmonary complications. Stroke. 2005 Dec;36(12):2756-63. doi: 10.1161/01.STR.0000190056.76543.eb. Epub 2005 Nov 3. PMID 16269630
- [Background] Ojo O, Brooke J. The Use of Enteral Nutrition in the Management of Stroke. Nutrients. 2016 Dec 20;8(12):827. doi: 10.3390/nu8120827. PMID 27999383
- [Background] Crary MA, Humphrey JL, Carnaby-Mann G, Sambandam R, Miller L, Silliman S. Dysphagia, nutrition, and hydration in ischemic stroke patients at admission and discharge from acute care. Dysphagia. 2013 Mar;28(1):69-76. doi: 10.1007/s00455-012-9414-0. Epub 2012 Jun 9. PMID 22684924
- [Background] Krekeler BN, Rowe LM, Connor NP. Dose in Exercise-Based Dysphagia Therapies: A Scoping Review. Dysphagia. 2021 Feb;36(1):1-32. doi: 10.1007/s00455-020-10104-3. Epub 2020 Mar 5. PMID 32140905
- [Background] McKenna VS, Zhang B, Haines MB, Kelchner LN. A Systematic Review of Isometric Lingual Strength-Training Programs in Adults With and Without Dysphagia. Am J Speech Lang Pathol. 2017 May 17;26(2):524-539. doi: 10.1044/2016_AJSLP-15-0051. PMID 28282484
- [Background] Smaoui S, Langridge A, Steele CM. The Effect of Lingual Resistance Training Interventions on Adult Swallow Function: A Systematic Review. Dysphagia. 2020 Oct;35(5):745-761. doi: 10.1007/s00455-019-10066-1. Epub 2019 Oct 14. PMID 31612288
- [Background] Moon JH, Hahm SC, Won YS, Cho HY. The effects of tongue pressure strength and accuracy training on tongue pressure strength, swallowing function, and quality of life in subacute stroke patients with dysphagia: a preliminary randomized clinical trial. Int J Rehabil Res. 2018 Sep;41(3):204-210. doi: 10.1097/MRR.0000000000000282. PMID 29621048
- [Background] Park JS, Kim HJ, Oh DH. Effect of tongue strength training using the Iowa Oral Performance Instrument in stroke patients with dysphagia. J Phys Ther Sci. 2015 Dec;27(12):3631-4. doi: 10.1589/jpts.27.3631. Epub 2015 Dec 28. PMID 26834320
- [Background] Steele CM, Bayley MT, Peladeau-Pigeon M, Nagy A, Namasivayam AM, Stokely SL, Wolkin T. A Randomized Trial Comparing Two Tongue-Pressure Resistance Training Protocols for Post-Stroke Dysphagia. Dysphagia. 2016 Jun;31(3):452-61. doi: 10.1007/s00455-016-9699-5. Epub 2016 Mar 2. PMID 26936446
- [Background] Steele CM, Cichero JA. Physiological factors related to aspiration risk: a systematic review. Dysphagia. 2014 Jun;29(3):295-304. doi: 10.1007/s00455-014-9516-y. Epub 2014 Feb 23. PMID 24562507
- [Background] McConnel FM. Analysis of pressure generation and bolus transit during pharyngeal swallowing. Laryngoscope. 1988 Jan;98(1):71-8. doi: 10.1288/00005537-198801000-00015. PMID 3336265
- [Background] Nicosia MA, Hind JA, Roecker EB, Carnes M, Doyle J, Dengel GA, Robbins J. Age effects on the temporal evolution of isometric and swallowing pressure. J Gerontol A Biol Sci Med Sci. 2000 Nov;55(11):M634-40. doi: 10.1093/gerona/55.11.m634. PMID 11078092
- [Background] Nicosia MA, Robbins JA. The fluid mechanics of bolus ejection from the oral cavity. J Biomech. 2001 Dec;34(12):1537-44. doi: 10.1016/s0021-9290(01)00147-6. PMID 11716855
- [Background] Clark HM. Neuromuscular treatments for speech and swallowing: a tutorial. Am J Speech Lang Pathol. 2003 Nov;12(4):400-15. doi: 10.1044/1058-0360(2003/086). PMID 14658992
- [Background] Todd JT, Lintzenich CR, Butler SG. Isometric and swallowing tongue strength in healthy adults. Laryngoscope. 2013 Oct;123(10):2469-73. doi: 10.1002/lary.23852. Epub 2013 Aug 5. PMID 23918664
- [Background] Kays SA, Hind JA, Gangnon RE, Robbins J. Effects of dining on tongue endurance and swallowing-related outcomes. J Speech Lang Hear Res. 2010 Aug;53(4):898-907. doi: 10.1044/1092-4388(2009/09-0048). PMID 20689047
- [Background] Clark HM. Specificity of training in the lingual musculature. J Speech Lang Hear Res. 2012 Apr;55(2):657-67. doi: 10.1044/1092-4388(2011/11-0045). Epub 2012 Jan 3. PMID 22215031
- [Background] Smithard DG, O'Neill PA, Parks C, Morris J. Complications and outcome after acute stroke. Does dysphagia matter? Stroke. 1996 Jul;27(7):1200-4. doi: 10.1161/01.str.27.7.1200. PMID 8685928
- [Background] Arnold M, Liesirova K, Broeg-Morvay A, Meisterernst J, Schlager M, Mono ML, El-Koussy M, Kagi G, Jung S, Sarikaya H. Dysphagia in Acute Stroke: Incidence, Burden and Impact on Clinical Outcome. PLoS One. 2016 Feb 10;11(2):e0148424. doi: 10.1371/journal.pone.0148424. eCollection 2016. PMID 26863627
- [Background] Patel DA, Krishnaswami S, Steger E, Conover E, Vaezi MF, Ciucci MR, Francis DO. Economic and survival burden of dysphagia among inpatients in the United States. Dis Esophagus. 2018 Jan 1;31(1):1-7. doi: 10.1093/dote/dox131. PMID 29155982
- [Background] Eslick GD, Talley NJ. Dysphagia: epidemiology, risk factors and impact on quality of life--a population-based study. Aliment Pharmacol Ther. 2008 May;27(10):971-9. doi: 10.1111/j.1365-2036.2008.03664.x. Epub 2008 Feb 28. PMID 18315591
- [Background] Robbins J, Kays SA, Gangnon RE, Hind JA, Hewitt AL, Gentry LR, Taylor AJ. The effects of lingual exercise in stroke patients with dysphagia. Arch Phys Med Rehabil. 2007 Feb;88(2):150-8. doi: 10.1016/j.apmr.2006.11.002. PMID 17270511
- [Background] Luker JA, Wall K, Bernhardt J, Edwards I, Grimmer-Somers K. Measuring the quality of dysphagia management practices following stroke: a systematic review. Int J Stroke. 2010 Dec;5(6):466-76. doi: 10.1111/j.1747-4949.2010.00488.x. PMID 21050403
- [Background] Geeganage C, Beavan J, Ellender S, Bath PM. Interventions for dysphagia and nutritional support in acute and subacute stroke. Cochrane Database Syst Rev. 2012 Oct 17;10:CD000323. doi: 10.1002/14651858.CD000323.pub2. PMID 23076886
- [Background] Rofes L, Vilardell N, Clave P. Post-stroke dysphagia: progress at last. Neurogastroenterol Motil. 2013 Apr;25(4):278-82. doi: 10.1111/nmo.12112. Epub 2013 Mar 11. PMID 23480388
- [Background] Cohen DL, Roffe C, Beavan J, Blackett B, Fairfield CA, Hamdy S, Havard D, McFarlane M, McLauglin C, Randall M, Robson K, Scutt P, Smith C, Smithard D, Sprigg N, Warusevitane A, Watkins C, Woodhouse L, Bath PM. Post-stroke dysphagia: A review and design considerations for future trials. Int J Stroke. 2016 Jun;11(4):399-411. doi: 10.1177/1747493016639057. Epub 2016 Mar 22. PMID 27006423
- [Background] Langmore SE, Pisegna JM. Efficacy of exercises to rehabilitate dysphagia: A critique of the literature. Int J Speech Lang Pathol. 2015 Jun;17(3):222-9. doi: 10.3109/17549507.2015.1024171. Epub 2015 Mar 31. PMID 25825989
- [Background] Swan K, Speyer R, Heijnen BJ, Wagg B, Cordier R. Living with oropharyngeal dysphagia: effects of bolus modification on health-related quality of life--a systematic review. Qual Life Res. 2015 Oct;24(10):2447-56. doi: 10.1007/s11136-015-0990-y. Epub 2015 Apr 14. PMID 25869989
- [Background] Rogus-Pulia N, Robbins J. Approaches to the rehabilitation of dysphagia in acute poststroke patients. Semin Speech Lang. 2013 Aug;34(3):154-69. doi: 10.1055/s-0033-1358368. Epub 2013 Oct 28. PMID 24166190
- [Background] Cullins MJ, Krekeler BN, Connor NP. Differential impact of tongue exercise on intrinsic lingual muscles. Laryngoscope. 2018 Oct;128(10):2245-2251. doi: 10.1002/lary.27044. Epub 2017 Dec 15. PMID 29243257
- [Background] Krekeler BN, Weycker JM, Connor NP. Effects of Tongue Exercise Frequency on Tongue Muscle Biology and Swallowing Physiology in a Rat Model. Dysphagia. 2020 Dec;35(6):918-934. doi: 10.1007/s00455-020-10105-2. Epub 2020 Mar 4. PMID 32130514
- [Background] Daniels SK, Brailey K, Foundas AL. Lingual discoordination and dysphagia following acute stroke: analyses of lesion localization. Dysphagia. 1999 Spring;14(2):85-92. doi: 10.1007/PL00009592. PMID 10028038
- [Background] Lee JH, Kim HS, Yun DH, Chon J, Han YJ, Yoo SD, Kim DH, Lee SA, Joo HI, Park JS, Kim JC, Soh Y. The Relationship Between Tongue Pressure and Oral Dysphagia in Stroke Patients. Ann Rehabil Med. 2016 Aug;40(4):620-8. doi: 10.5535/arm.2016.40.4.620. Epub 2016 Aug 24. PMID 27606268
- [Background] Crary MA, Mann GD, Groher ME. Initial psychometric assessment of a functional oral intake scale for dysphagia in stroke patients. Arch Phys Med Rehabil. 2005 Aug;86(8):1516-20. doi: 10.1016/j.apmr.2004.11.049. PMID 16084801
- [Background] Martin-Harris B, Brodsky MB, Michel Y, Castell DO, Schleicher M, Sandidge J, Maxwell R, Blair J. MBS measurement tool for swallow impairment--MBSImp: establishing a standard. Dysphagia. 2008 Dec;23(4):392-405. doi: 10.1007/s00455-008-9185-9. Epub 2008 Oct 15. PMID 18855050
- [Background] Beall J, Hill EG, Armeson K, Garand KLF, Davidson KH, Martin-Harris B. Classification of Physiologic Swallowing Impairment Severity: A Latent Class Analysis of Modified Barium Swallow Impairment Profile Scores. Am J Speech Lang Pathol. 2020 Jul 10;29(2S):1001-1011. doi: 10.1044/2020_AJSLP-19-00080. Epub 2020 Jul 10. PMID 32650665
- [Background] Martin-Harris B, Garand KLF, McFarland D. Optimizing Respiratory-Swallowing Coordination in Patients With Oropharyngeal Head and Neck Cancer. Perspect ASHA Spec Interest Groups. 2017 Jul;2(13):103-110. doi: 10.1044/persp2.SIG13.103. Epub 2017 Jul 31. PMID 28884146
- [Background] Pearson WG Jr, Molfenter SM, Smith ZM, Steele CM. Image-based measurement of post-swallow residue: the normalized residue ratio scale. Dysphagia. 2013 Jun;28(2):167-77. doi: 10.1007/s00455-012-9426-9. Epub 2012 Oct 23. PMID 23089830
- [Background] Rosenbek JC, Robbins JA, Roecker EB, Coyle JL, Wood JL. A penetration-aspiration scale. Dysphagia. 1996 Spring;11(2):93-8. doi: 10.1007/BF00417897. PMID 8721066
- [Background] Carnaby-Mann GD, Crary MA. Adjunctive neuromuscular electrical stimulation for treatment-refractory dysphagia. Ann Otol Rhinol Laryngol. 2008 Apr;117(4):279-87. doi: 10.1177/000348940811700407. PMID 18478837
- [Background] Schneider CA, Rasband WS, Eliceiri KW. NIH Image to ImageJ: 25 years of image analysis. Nat Methods. 2012 Jul;9(7):671-5. doi: 10.1038/nmeth.2089. PMID 22930834
- [Background] Robbins J, Coyle J, Rosenbek J, Roecker E, Wood J. Differentiation of normal and abnormal airway protection during swallowing using the penetration-aspiration scale. Dysphagia. 1999 Fall;14(4):228-32. doi: 10.1007/PL00009610. PMID 10467048
- [Background] Steele CM, Grace-Martin K. Reflections on Clinical and Statistical Use of the Penetration-Aspiration Scale. Dysphagia. 2017 Oct;32(5):601-616. doi: 10.1007/s00455-017-9809-z. Epub 2017 May 22. PMID 28534064
- [Background] Bonilha HS, Wilmskoetter J, Tipnis SV, Martin-Harris B, Huda W. EFFECTIVE DOSE PER UNIT KERMA-AREA PRODUCT CONVERSION FACTORS IN ADULTS UNDERGOING MODIFIED BARIUM SWALLOW STUDIES. Radiat Prot Dosimetry. 2017 Nov 1;176(3):269-277. doi: 10.1093/rpd/ncx006. PMID 28204745
- [Background] Bonilha HS, Huda W, Wilmskoetter J, Martin-Harris B, Tipnis SV. Radiation Risks to Adult Patients Undergoing Modified Barium Swallow Studies. Dysphagia. 2019 Dec;34(6):922-929. doi: 10.1007/s00455-019-09993-w. Epub 2019 Mar 4. PMID 30830303
- [Background] Hendee WR, Edwards FM. ALARA and an integrated approach to radiation protection. Semin Nucl Med. 1986 Apr;16(2):142-50. doi: 10.1016/s0001-2998(86)80027-7. PMID 3961515
- [Background] Fullerton HJ, Wu YW, Zhao S, Johnston SC. Risk of stroke in children: ethnic and gender disparities. Neurology. 2003 Jul 22;61(2):189-94. doi: 10.1212/01.wnl.0000078894.79866.95. PMID 12874397
- [Background] Bigi S, Fischer U, Wehrli E, Mattle HP, Boltshauser E, Burki S, Jeannet PY, Fluss J, Weber P, Nedeltchev K, El-Koussy M, Steinlin M, Arnold M. Acute ischemic stroke in children versus young adults. Ann Neurol. 2011 Aug;70(2):245-54. doi: 10.1002/ana.22427. PMID 21823153

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lingual Endurance Training
Started | 19
Completed | 15
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- Lingual Endurance Training: Intervention group will complete lingual endurance training. Half of the participants also completed effortful swallows once per day
  Lingual Endurance Exercise: Participants will participate in 3 training sessions per day for 8 weeks. Half of the participants completed 3 sessions of lingual endurance exercise. For example, if the participant completed 100 repetitions during the baseline measurement, they would complete 75 repetitions during their exercise session. The other half completed 2 of these sessions, with 1 session of effortful swallow practice (10 repetitions)
Arm/Group | Lingual Endurance Training
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Adherence
Description: % [(total number of days of attempted exercise/total number of days prescribed over 8 weeks of therapy)x100]
Time Frame: Assessed at 8 weeks (study completion)
Population: Only participants that completed baseline and final visits
Measure: Mean (Standard Deviation); unit: percentage of adherence
Arm/Group | Lingual Endurance Training
Number analyzed (Participants) | 15
percentage of adherence | 79 (29)

2. Primary Outcome: Change From Baseline Modified Barium Swallowing Impairment Profile (MBSImP) Oral Total Score
Description: Improvement on Oral Total (OT) score MBSImP; OT score minimum score (best) =0; OT maximum score (worst) = 22
Time Frame: Baseline and 8 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lingual Endurance Training
Number analyzed (Participants) | 15
score on a scale | 0.2667 (2.82)
Statistical Analysis 1: Comparison: Lingual Endurance Training; Test type: Superiority; p = 0.66, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Participant Improving Worst Penetration Aspiration Scale (PAS) Score
Description: measure of airway invasion during swallowing, best score = 1, worst score = 8 Number of patients who improved worst PAS score from baseline to 8 week timepoint
Time Frame: Baseline and 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lingual Endurance Training
Number analyzed (Participants) | 15
Participants | 6
Statistical Analysis 1: Comparison: Lingual Endurance Training; Test type: Superiority; p = 1.0, Chi-squared

4. Secondary Outcome: Change From Baseline in Post-swallow Residue (Solid)
Description: Analysis of Swallowing Physiology, Kinematics, Events, Timing (ASPEKT): The ASPEKT method uses ImageJ pixel based measures of post-swallow residue (Total% of C2-C4)
Time Frame: Baseline and 8 Weeks
Measure: Mean (Standard Deviation); unit: percent of C2-C4
Arm/Group | Lingual Endurance Training
Number analyzed (Participants) | 15
percent of C2-C4 | -1.33 (2.5)
Statistical Analysis 1: Comparison: Lingual Endurance Training; Test type: Superiority; p = 0.09, Sign test

5. Secondary Outcome: Change From Baseline in Post-swallow Residue (Puree)
Description: as for outcome 4
Time Frame: Baseline and 8 Weeks
Measure: Mean (Standard Deviation); unit: percent of C2-C4
Arm/Group | Lingual Endurance Training
Number analyzed (Participants) | 15
percent of C2-C4 | -.67 (6.6)
Statistical Analysis 1: Comparison: Lingual Endurance Training; Test type: Superiority; p = .722, Sign test

6. Secondary Outcome: Change From Baseline in Post-swallow Residue (Thin Liquids)
Description: as for outcome 4
Time Frame: Baseline and 8 Weeks
Measure: Mean (Standard Deviation); unit: percent of C2-C4
Arm/Group | Lingual Endurance Training
Number analyzed (Participants) | 10
percent of C2-C4 | -1.5 (4.2)
Statistical Analysis 1: Comparison: Lingual Endurance Training; Test type: Superiority; p = .28, Sign test

7. Secondary Outcome: Change From Baseline in Post-swallow Residue (Mildly Thick Liquids)
Description: as for outcome 4
Time Frame: Baseline and 8 Weeks
Measure: Mean (Standard Deviation); unit: percent of C2-C4
Arm/Group | Lingual Endurance Training
Number analyzed (Participants) | 11
percent of C2-C4 | -1.01 (2.58)
Statistical Analysis 1: Comparison: Lingual Endurance Training; Test type: Superiority; p = .15, Sign test

8. Secondary Outcome: Change From Baseline in Post-swallow Residue (Moderately Thick Liquids)
Description: as for outcome 4
Time Frame: Baseline and 8 Weeks
Measure: Mean (Standard Deviation); unit: percent of C2-C4
Arm/Group | Lingual Endurance Training
Number analyzed (Participants) | 14
percent of C2-C4 | .25 (5.0)
Statistical Analysis 1: Comparison: Lingual Endurance Training; Test type: Superiority; p = .8, Sign test

9. Secondary Outcome: Change From Baseline in Swallowing Quality of Life Questionnaire (SWAL-QoL)
Description: Patient reported outcome measure of swallowing quality of life, 0 = best score; 100 = worst score
Time Frame: Baseline and 8 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lingual Endurance Training
Number analyzed (Participants) | 14
score on a scale | 8.3 (18.74)
Statistical Analysis 1: Comparison: Lingual Endurance Training; Test type: Superiority; p = .12, t-test, 2 sided

10. Secondary Outcome: Change From Baseline Eating Assessment Tool (EAT-10) Score
Description: patient reported outcome tool; 0 = best score, 50 = worst score
Time Frame: Baseline and 8 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lingual Endurance Training
Number analyzed (Participants) | 15
score on a scale | -0.0667 (4.93)
Statistical Analysis 1: Comparison: Lingual Endurance Training; Test type: Superiority; p = .92, Sign test

ADVERSE EVENTS:
Time Frame: Participants were enrolled on average 8-10 weeks
Description: Only 2 participants were hospitalized due to non-protocol related reasons
Arm/Group | Lingual Endurance Training
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 2/19
Other Adverse Events (participants affected / at risk) | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lingual Endurance Training (N=19)
Hospitalization (Infections and infestations) | 2 (2) — 2 patients hospitalized due to non-study related infections (pneumonia)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-18): https://cdn.clinicaltrials.gov/large-docs/73/NCT05523973/Prot_SAP_000.pdf